CLINICAL TRIAL: NCT04912726
Title: Efficacy and Safety of Endovenous Sildenafil Early Management in Newborns Pulmonary Hypertension: a Clinical Trial
Brief Title: Endovenous Sildenafil Early Management in Newborns Pulmonary Hypertension
Acronym: HIPSEN
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study did not begin due to lack of resources for its execution.
Sponsor: Universidad del Norte (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 234
Record Dates: First submitted 2021-05-24; First posted 2021-06-03 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Hypertension, Pulmonary
Keywords: newborn; intravenous sildenafil; Hypertension, Pulmonary
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, double-blind clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Assignment concealment will be ensured using sealed and sequenced opaque (dark) sealed envelopes containing the assignments. An investigator will carry out the assignment, write down the assignment number in a specific format, seal the opaque envelope and number it consecutively. These envelopes will be stored in the neonatal intensive care unit of the hospital child jesus where the study will be carried out. Once a subject has met the inclusion criteria, the neonatal intensive care unit pharmacy service will be notified, staff not participating in the study who will make a phone call to the investigator so that he can assign the label number to the new subject who I enter the study, the pharmacy shift personnel are in charge of labeling and delivering the product to the nursing staff. The active product intravenous sildenafil and the placebo are packaged in identical burette, the burette content is visible and the coloration is transparent.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive intravenous sildenafil loading dose of 0.4 mg / kg in 3 hours and continue in continuous infusion at 1.6 mg / kg / day (0.067 mg / kg / h).
  Interventions: Drug: Sildenafil Injectable Product
- Placebo (No Intervention): The control group will receive placebo at the same loading dose and infusion with 0.9% saline solution plus standard management under the unit protocol immediately after the echocardiographic diagnosis.

INTERVENTIONS:
Drug: Sildenafil Injectable Product — The intervention group will receive intravenous sildenafil loading dose of 0.4 mg / kg in 3 hours and continue in continuous infusion at 1.6 mg / kg / day (0.067 mg / kg / h).
  Other Names: Intravenous sildenafil
  Arms: Intervention

SUMMARY:
Sildenafil is currently approved for the management of pulmonary hypertension of the newborn, with the availability of intravenous presentation it has been seen that the severity condition has already established, many times these patients do not have the adequate clinical response and there are no studies to date that evaluate the efficacy and safety of the same when it is started early in these patients, therefore we plan a randomized clinical trial to determine the efficacy and safety of the administration of intravenous sildenafil for early management of newborns with persistent pulmonary hypertension of the newborn.

DETAILED DESCRIPTION:
Persistent pulmonary hypertension of the newborn is a relatively common condition that occurs in 2 to 7/1000 live births, being higher in term and late preterm newborns, representing up to 4% of all admissions in some units neonatal intensive care and that results in a mortality that ranges between 4 and 33% in the world. In the United States, its incidence varies between 0.4 and 6.8 per 1000 live births, while in the United Kingdom it is between 0.43 and 6 per 1000 live births. Although there has been an important development in the treatment of persistent pulmonary hypertension of the newborn in the last time, its impact on early neonatal mortality continues to be important, reaching approximately 10%. Currently there are no mortality data in underdeveloped countries and in Latin America. This considerable mortality is most likely a consequence of the fact that 40% of newborns are resistant to inhaled nitric oxide, which, together with supportive therapies, is the basis of treatment. Furthermore, the increasing cost of administering Nitric oxide to infants with pulmonary hypertension of the newborn reduces its availability in developing countries. On the other hand, extracorporeal membrane oxygenation is another therapeutic option that is currently being systematically evaluated in clinical trials, even so, it is not available in all units. Therefore, there was a real need to evaluate novel approaches for the management of the disease, being necessary to create therapeutic strategies that allow improving the prognosis of these newborns. Sildenafil is currently approved for the management of persistent pulmonary hypertension of the newborn, with the availability of intravenous presentation it has been seen that once the severity picture has been established, many times these patients do not have the adequate clinical response and there are no studies to date that evaluate the efficacy and safety of the same when started early in these patients.

Primary outcome: To assess the efficacy in decreasing estimated pulmonary artery pressure by 20% and improving survival with early use of intravenous sildenafil at a loading dose of 0.4 mg / kg in 3 hours, followed of continuous infusion at 1.6 mg / kg / day versus conventional treatment plus placebo in neonates with persistent pulmonary hypertension of the newborn.

Materials and methods:

A total of 44 newborns with a gestational age ≥ 34 weeks of age and less than 10 days old who were admitted to the Neonatal Intensive Care Unit, High Complexity Medicine with a diagnosis of persistent pulmonary hypertension of the newborn in absentia, were evaluated. of congenital heart disease or oxygenation index greater than 15, attended between May 2021 and May 2022 in the city of Barranquilla, 22 were divided into two groups for the control group and 22 for the intervention group. the intervention group received intravenous sildenafil loading dose of 0.4 mg / kg in 3 hours and continued in continuous infusion at 1.6 mg / kg / day (0.067 mg / kg / h). The control group will receive placebo at the same loading dose and infusion with 0.9% saline solution plus standard management under the unit protocol immediately after the echocardiographic diagnosis. The measure of the primary outcome was given by the decrease of 20% in the estimated pressure of the pulmonary artery by echocardiography at 24 hours after the start of treatment, at 48 hours, between 96 - 168 hours and 48 hours after the drug discontinuation.

Results and conclusions: ongoing.

Declaration of conflict of interest: The authors do not present any situation of real, potential or evident conflict of interest, including any financial or other interest.

ELIGIBILITY:
Inclusion Criteria:

* Newborns with gestational age ≥ 34 weeks and less than 10 days old, from the delivery room, joint accommodation, surgery at the Niño Jesus Hospital and referred from other institutions with an echocardiographic diagnosis of persistent pulmonary hypertension of the newborn. A diagnosis of persistent pulmonary hypertension of the newborn will be made if any of the following criteria are identified in the absence of cyanotic congenital heart disease by echocardiography: Tricuspid regurgitant jet with a pressure gradient ≥ 2/3 of systemic systolic blood pressure; intraventricular septum that flattens or slopes into the left ventricular cavity; bidirectional or right-to-left flow through patent ductus arteriosus; pulmonary artery acceleration time <40 milliseconds

Exclusion Criteria:

* Congenital heart disease or fatal congenital anomalies
* Oxygenation Index (IO) > 15
* No parental consent

Max Age: 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
20% decrease in estimated pulmonary artery pressure | 7 days
  Evaluate the efficacy in lowering the estimated pulmonary artery pressure by 20% and improved survival with early use of intravenous sildenafil at a loading dose of 0.4 mg / kg in 3 hours, followed by continuous infusion at 1.6 mg / kg / day versus conventional treatment plus placebo in neonates with persistent pulmonary hypertension of the newborn.

SECONDARY OUTCOMES:
Duration of mechanical ventilation | 7 days
  Evaluate the duration of mechanical ventilation with early use of intravenous sildenafil at a loading dose of 0.4 mg / kg in 3 hours, followed by continuous infusion at 1.6 mg / kg / day versus conventional treatment plus placebo in neonates with persistent pulmonary hypertension of the newborn.
Duration of inotropic therapy | 7 days
  To assess the duration of inotropic therapy with early use of intravenous sildenafil at a loading dose of 0.4 mg / kg in 3 hours, followed by continuous infusion at 1.6 mg / kg / day versus conventional treatment. plus placebo in neonates with persistent pulmonary hypertension of the newborn.
Adverse events | 7 days
  Correlate the presence of adverse events such as arterial hypotension, the presence of bleeding and retinopathy of prematurity with the early use of intravenous sildenafil at a loading dose of 0.4 mg / kg in 3 hours, followed by continuous infusion at 1.6 mg / kg / day versus conventional treatment plus placebo in neonates with persistent pulmonary hypertension of the newborn.

REFERENCES:
- [Background] Martinho S, Adao R, Leite-Moreira AF, Bras-Silva C. Persistent Pulmonary Hypertension of the Newborn: Pathophysiological Mechanisms and Novel Therapeutic Approaches. Front Pediatr. 2020 Jul 24;8:342. doi: 10.3389/fped.2020.00342. eCollection 2020. PMID 32850518
- [Background] Jain A, McNamara PJ. Persistent pulmonary hypertension of the newborn: Advances in diagnosis and treatment. Semin Fetal Neonatal Med. 2015 Aug;20(4):262-71. doi: 10.1016/j.siny.2015.03.001. Epub 2015 Apr 2. PMID 25843770
- [Background] Fuloria M, Aschner JL. Persistent pulmonary hypertension of the newborn. Semin Fetal Neonatal Med. 2017 Aug;22(4):220-226. doi: 10.1016/j.siny.2017.03.004. Epub 2017 Mar 23. PMID 28342684
- [Background] Baquero H, Soliz A, Neira F, Venegas ME, Sola A. Oral sildenafil in infants with persistent pulmonary hypertension of the newborn: a pilot randomized blinded study. Pediatrics. 2006 Apr;117(4):1077-83. doi: 10.1542/peds.2005-0523. PMID 16585301
- [Background] Pedersen J, Hedegaard ER, Simonsen U, Kruger M, Infanger M, Grimm D. Current and Future Treatments for Persistent Pulmonary Hypertension in the Newborn. Basic Clin Pharmacol Toxicol. 2018 Oct;123(4):392-406. doi: 10.1111/bcpt.13051. Epub 2018 Jul 19. PMID 29855164
- [Background] Lakshminrusimha S, Mathew B, Leach CL. Pharmacologic strategies in neonatal pulmonary hypertension other than nitric oxide. Semin Perinatol. 2016 Apr;40(3):160-73. doi: 10.1053/j.semperi.2015.12.004. Epub 2016 Jan 14. PMID 26778236
- [Background] El-Khuffash A, McNamara PJ, Breatnach C, Bussmann N, Smith A, Feeney O, Tully E, Griffin J, de Boode WP, Cleary B, Franklin O, Dempsey E. The use of milrinone in neonates with persistent pulmonary hypertension of the newborn - a randomised controlled trial pilot study (MINT 1): study protocol and review of literature. Matern Health Neonatol Perinatol. 2018 Dec 3;4:24. doi: 10.1186/s40748-018-0093-1. eCollection 2018. PMID 30524749
- [Background] Uslu S, Kumtepe S, Bulbul A, Comert S, Bolat F, Nuhoglu A. A comparison of magnesium sulphate and sildenafil in the treatment of the newborns with persistent pulmonary hypertension: a randomized controlled trial. J Trop Pediatr. 2011 Aug;57(4):245-50. doi: 10.1093/tropej/fmq091. Epub 2010 Oct 4. PMID 20923790